CLINICAL TRIAL: NCT04052529
Title: Impact of Using Self-monitoring Smartphone Applications on College Students' Well-being
Brief Title: Tracking Our Lives Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Samantha Hahn, PhD Candidate, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00161687
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Mental Health Wellness 2; Health Behavior; Eating Disorders
MeSH Terms: conditions — Health Behavior; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants are instructed to use a popular dietary self-monitoring application on their smartphone for one month.
  Interventions: Other: Dietary self-monitoring
- Control (No Intervention): Participants are not asked to use the smartphone application.

INTERVENTIONS:
Other: Dietary self-monitoring — Participants use a popular smartphone application to track their food and drink intake for one month.
  Arms: Intervention

SUMMARY:
College women are at risk for eating disorders, which have profound health impacts. Cross-sectional studies have shown that the use of dietary self-monitoring is associated with eating disorder risk among college students. However, causality cannot be established with cross-sectional studies.

This study utilizes a randomized controlled trial design to examine how the use of a popular dietary self-monitoring smartphone application impacts college females' well-being, including eating disorder risk. We hypothesize those who are randomized to dietary self-monitoring will have a greater increase in eating disorder risk compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* University of Michigan Ann Arbor undergraduate student
* Daily access to a smartphone
* Female gender
* At least 18 years of age
* Fluent in English

Exclusion Criteria:

* Self-reported history of any medical condition that impacts the types or amount of food eaten
* Self-reported recent use of dietary self-monitoring
* Self-reported history of an active or past eating disorder
* Eating Disorder Examination Questionnaire Short Form (EDE-QS) score ≥ 2, indicating high eating disorder risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as female.
Enrollment: 200 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Risk | 30 days
  Eating disorder risk will be measured on a survey via the Eating Disorder Examination Questionnaire Short Form (EDE-QS). The EDE-QS is a validated 12 question scale. Each question has a score range 0-3, and the average of all scores is the overall score. A higher score indicates higher risk.
Eating Disorder Risk | 30 days
  Measured via survey using the validated SCOFF questionnaire which consists of five questions. Each question is a yes/no and a yes receives one point with a total score ranging from 0-5. Higher scores indicate higher risk. Modified to ask about pounds instead of stone as a measure of weight.

SECONDARY OUTCOMES:
Weight-Related Self-Monitoring | 30 days
  Measured via survey that includes single item measures asking about physical activity self-monitoring and self-weighing frequency.
Body Image | 30 days
  Assessed via survey using the validated 6 question Body Image States Scale (BISS). Scores are the mean of the six items, three of which are reverse coded. Higher scores mean better body image states.
Weight Stigma | 30 days
  Measured via survey using five single item questions.
Dietary Intake | 30 days
  Single item survey questions adapted from the Youth Risk Behavior Surveillance System
Physical Activity | 30 days
  Single item survey questions adapted from the Youth Risk Behavior Surveillance System and an open ended question for amount of time physically active.
Weight perception | 30 days
  Assessed using two questions on a survey pertaining to BMI category and weight.
Body changing intentions | 30 days
  Assessed using single item question on a survey asking how, if at all, participants wanted to change their body.
Social Media Use | 30 days
  Use of common social media sites assessed using five single item measures on a survey.
Weight | 30 days
  Blind weights taken on research grade laboratory scale.
Subjective Quality of Life | 30 days
  Assessed using the Brunnsviken Brief Quality of Life Scale (BBQ) on a survey. The BBQ has 12 questions, each ranging from 0-4. Higher scores indicate higher subjective quality of life.
Anxiety | 30 days
  State anxiety as measured via survey using the short-form of the state scale of the Spielberger State-Trait Anxiety Inventory. The scale consists of 6 questions with a range of scores 1-4 for each question. Three positive questions are reverse coded and scores are added together with higher scores indicating higher state anxiety.
Depression Symptoms | 30 days
  Measured via survey using the Center for Epidemiologic Studies Depression Scale Revised (CESD-R-10). The CESD-R-10 is a 10 item scale with each question having the possibility of a score 0-3. Two questions are reverse coded, then scores from each question are added to give an overall score. Higher scores indicate more depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Hahn SL, Kaciroti N, Eisenberg D, Weeks HM, Bauer KW, Sonneville KR. Introducing Dietary Self-Monitoring to Undergraduate Women via a Calorie Counting App Has No Effect on Mental Health or Health Behaviors: Results From a Randomized Controlled Trial. J Acad Nutr Diet. 2021 Dec;121(12):2377-2388. doi: 10.1016/j.jand.2021.06.311. Epub 2021 Aug 20. PMID 34427188